CLINICAL TRIAL: NCT01812096
Title: Prospective Comparison the Pharmacokinetics of Subcutaneous Versus Intravenous Administration of Bortezomib in Newly Diagnosed Patients of Multiple Myeloma in China.
Brief Title: Study of Subcutaneous Versus Intravenous Administration of Bortezomib in Patients With Multiple Myeloma in China
Acronym: MM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SZ5201
Record Dates: First submitted 2013-03-13; First posted 2013-03-15 (Estimated); Last update posted 2015-08-18 (Estimated); Status verified 2015-08

CONDITIONS: Multiple Myeloma Proved by Laboratory Tests
Keywords: multiple myeloma; bortezomib; Subcutaneous
MeSH Terms: conditions — Multiple Myeloma

ARMS (2):
- the pharmacokinetic of bortezomib (Experimental): the pharmacokinetic and pharmacodynamic, and assessed safety and efficacy of subcutaneous administration of bortezomib
  Interventions: Other: Subcutaneous bortezomib
- Intravenous (Active Comparator): the pharmacokinetic and pharmacodynamic, and assessed safety and efficacy of intravenous administration of bortezomib
  Interventions: Other: Intravenous bortezomib

INTERVENTIONS:
Other: Subcutaneous bortezomib
  Other Names: the methods of use bortezomib
  Arms: the pharmacokinetic of bortezomib
Other: Intravenous bortezomib
  Arms: Intravenous

SUMMARY:
Intravenous injection is the standard administration route of bortezomib; however, subcutaneous administration is an important alternative. We want to compared the pharmacokinetic of subcutaneous versus intravenous bortezomib at the approved 1•3 mg/m2 dose and twice per week,on days1, 4, 8 and 11 of 21-day cycles, schedule in newly diagnosed patients of multiple myeloma.

DETAILED DESCRIPTION:
The new diagnosed multiple myeloma patients are randomized to receive bortezomib by standard intravenous bolus (n=10) or subcutaneous injection (n=10) at the recommended dose and schedule (1.3 mg/m2), days 1, 4, 8, 11;eight 21-day cycles).

Patients discontinued treatment due to progressive disease, insufficient efficacy, unacceptable toxicity, or serious protocol violation. Dose modifications are specified for unexpected pharmacokinetic observations or toxicity. Bortezomib-related neuropathic pain and/or peripheral sensory neuropathy were managed using established dose-modification guidelines.

Blood samples for pharmacokinetic/pharmacodynamic analysis are collected on days 1 and 11, cycle 1:before bortezomib administration, and at 2, 5, 15, 30, and 60 min, and 2, 4, 6, 10, 24, 32, 48, and 72 hours post-dosing. Pharmacodynamic analyses were performed using a whole-blood 20S proteasome specific activity inhibition assay.

ELIGIBILITY:
Inclusion Criteria:

* Must be Multiple Myeloma Proved by Laboratory Tests
* Must have the ability to observe the efficacy and events
* Patient must have the ability to understand and willingness to provide written informed consent in the study and any related procedures being performed

Exclusion Criteria:

* If have uncontrolled intercurrent illness including ongoing or active infection,heart failure,unstable angina pectoris,or psychiatric illness/social situations that study requirements
* If have severe side-effects on bortezomib

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-05; Primary Completion 2016-01 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
pharmacokinetic | 6 months

SECONDARY OUTCOMES:
curative effect | two years

CONTACTS AND LOCATIONS:
Overall Officials: Fu chengcheng, PhD, Principal Investigator — First Affiliated Hospital,Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China